CLINICAL TRIAL: NCT05561426
Title: Sustained Effect of Food Texture of Ultra-processed Foods on Energy Intake
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wageningen University (Other)
Responsible Party: Principal Investigator, Ciaran Forde, prof.dr. CG (Ciarán) Forde, Wageningen University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: PRESTRUCTURE
Record Dates: First submitted 2022-09-20; First posted 2022-09-30 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Eating Behavior
Keywords: Food texture; Ultra-processed foods; Food intake; Energy intake; Eating rate
MeSH Terms: conditions — Feeding Behavior

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fast UPF meals (Experimental): Meals consisting of UPF with textures that are consumed fast
  Interventions: Other: Ad libitum breakfast and dinner meals for 12 days
- Slow UPF meals (Experimental): Meals consisting of UPF with textures that are consumed slow
  Interventions: Other: Ad libitum breakfast and dinner meals for 12 days

INTERVENTIONS:
Other: Ad libitum breakfast and dinner meals for 12 days — Ad libitum portions of breakfast and dinner meals served at the eating behaviour lab

SUMMARY:
In this study the sustained effect of food texture differences (slow vs fast eating rate) of ultra-processed foods on energy intake and body composition changes will be investigated.

DETAILED DESCRIPTION:
Rationale: Several observational studies have shown that the consumption of ultra-processed foods (UPF) is associated with higher energy intake and obesity rates. However, the high eating rate of UPF might cause its high energy intake instead of the industrial processing level itself. There is a positive relationship between the eating rate and oro-sensory exposure of foods and subsequent energy intake. Food texture modifies eating rate and through that the energy intake of foods. It is shown that harder, chunkier, more viscous, and more voluminous foods decrease eating rate of foods and thus decrease energy intake. So far, research on food texture and energy intake has only been performed for one meal or one day and it is unknown if food texture and eating rate have a sustained effect on energy intake. Knowledge on the sustained effect of food texture differences could be used for strategies to drive or limit energy intake.

Objective: The primary objective is to determine the sustained effect of food texture differences (slow vs fast eating rate) of UPF on energy intake. The secondary objective is to determine the effect of texture differences (slow vs fast eating rate) of UPF on body composition changes.

Study design: The study has a randomized crossover design with two treatment arms. All participants receive both conditions (1. slow test breakfast and dinners consisting of UPF and 2. fast test breakfast and dinners consisting of UPF for twelve subsequent days) and are their own control (within subject effects).

Study population: Healthy Dutch speaking adults (n=20) between 18-55 years old with a BMI between 18.5-30 kg/m2.

Intervention: Participants will join two test periods, each consisting out of twelve days. During the test periods they will visit the eating behaviour lab where they receive ad libitum breakfast and dinner meals. During meal consumption participants are video recorded to determine eating behaviour. Standardized fixed portion lunch meals and snacks will be provided on-the-go. On weekend days participants will receive pre-packed meals. In one test period participants will receive meals consisting of UPF that have a hard texture (slow eating rate) and in the other period (randomized order) they will receive meals consisting of UPF with a soft texture (fast eating rate). The order in which participants will receive the meals within each condition will be (block) randomized.

ELIGIBILITY:
Inclusion Criteria:

* Between 18-55 years old at the day of inclusion
* Able to understand and speak Dutch and English fluently or without difficulty (self-report)
* BMI 18.5-30 kg/m2 - measured by the researchers during the information meeting (after signing informed consent)
* Good general health and appetite (self-report)
* Commonly (5 out of 7 week days) eating three meals a day every day around approximately the same times (self-report)

Exclusion Criteria:

* Difficulties with swallowing, chewing, and/or eating in general
* Suffering from an endocrine or eating disorder, gastrointestinal illness or illness of the thyroid gland, respiratory disease, or diabetes
* Having taste or smell disorders (self-report)
* Braces (not including a dental wire) or oral piercing
* Smoking
* Consuming on average more than 21 glasses of alcohol per week
* Not willing to stop using drugs during the study period (from inclusion till last test session)
* Use of medication that may influence study outcomes (self-report)
* Allergies or intolerance to any ingredient of the test meals
* Not willing to eat the test food because of eating habits, believes, or religion
* Following a vegetarian or vegan diet
* Lactose intolerant
* Men having facial hair such as a beard as facial movements cannot be analysed
* Followed an energy restricted diet during the last 2 months
* Gained or lost 5 kg of body weight over the last half year
* High restrained eater according to the Dutch Eating Behaviour Questionnaire (men: score>2.89, women>3.39) - this exclusion criterion will not explicitly be communicated to the participants to prevent desirable answers
* Signed up for participating in another research study of the Nutrition and Health department (WUR)
* Employee, thesis student or intern at the chair group of Sensory Science and Eating Behaviour Human Nutrition (WUR).
* Intensive exercising more than 5 hours per week
* Low score (<1) for liking the individual test meals on a nine point Likert scale based on pictures of the meals
* Unfamiliar with the test meals (self-report)
* Having an abnormal (non-representative) eating rates - measured by the researchers during the information meeting (after signing informed consent)

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2023-02-13 (Actual); Primary Completion 2023-04-14 (Actual); Study Completion 2023-04-14 (Actual)

PRIMARY OUTCOMES:
Average daily energy intake (kcal/day) | Two periods of 12 days
  Daily energy intake across 12 days for each diet

SECONDARY OUTCOMES:
Body weight (kg) | Two periods of 12 days
  Body weight (kg) measured using in duplicate using a weighing scale
Fat free mass measured with bioelectrical impedance analysis | Two periods of 12 days
  Fat free mass measured with bioelectrical impedance analysis (kg and %)
Fat free mass measured with skinfold measurements | Two periods of 12 days
  Fat free mass measured with skinfold measurements (kg and %)
Fat mass measured with bioelectrical impedance analysis | Two periods of 12 days
  Fat mass measured wit bioelectrical impedance analysis (kg and %)
Fat mass measured with skinfold measurements | Two periods of 12 days
  Fat mass measured with skinfold measurements (kg and %)
Waist and hip circumference (cm) | Two periods of 12 days
  Waist and hip circumference will be measured in duplicate using measuring tape
BMI | Two periods of 12 days
  Obtained by body weight (kg; measured using a weighing scale) and height (cm; measured using a stadiometer)

OTHER OUTCOMES:
Subjective hunger | Two periods of 12 days
  Hunger measured before and 0, 30, 60 and 90 minutes after meal consumption on a 100-mm VAS ranging from 'not at all' (0) to 'extremely' (100) with anchors at the beginning and end of the line
Subjective fullness | Two periods of 12 days
  Fullness measured before and 0, 30, 60 and 90 minutes after meal consumption on a 100-mm VAS ranging from 'not at all' (0) to 'extremely' (100) with anchors at the beginning and end of the line
Subjective desire to eat | Two periods of 12 days
  Desire to eat measured before and 0, 30, 60 and 90 minutes after meal consumption on a 100-mm VAS ranging from 'not at all' (0) to 'extremely' (100) with anchors at the beginning and end of the line
Subjective prospective consumption | Two periods of 12 days
  Prospective consumption measured before and 0, 30, 60 and 90 minutes after meal consumption on a 100-mm VAS ranging from 'not at all' (0) to 'extremely' (100) with anchors at the beginning and end of the line
Liking | Two periods of 12 days
  Liking of meals after one bite and after meal consumption will be rated on a 100-mm VAS scale ranging from 'not at all' to 'extremely' with anchors at the beginning and end of the line
Flavour intensity | Two periods of 12 days
  Flavour intensity after one bite will be rated on a 100-mm VAS scale ranging from 'not at all' to 'extremely' with anchors at the beginning and end of the line
Sweetness | Two periods of 12 days
  Sweetness intensity after one bite will be rated on a 100-mm VAS scale ranging from 'not at all' to 'extremely' with anchors at the beginning and end of the line
Sourness | Two periods of 12 days
  Sourness intensity after one bite will be rated on a 100-mm VAS scale ranging from 'not at all' to 'extremely' with anchors at the beginning and end of the line
Saltiness | Two periods of 12 days
  Saltiness intensity after one bite will be rated on a 100-mm VAS scale ranging from 'not at all' to 'extremely' with anchors at the beginning and end of the line
Hardness | Two periods of 12 days
  Hardness after one bite will be rated on a 100-mm VAS scale ranging from 'not at all' to 'extremely' with anchors at the beginning and end of the line
Firmness | Two periods of 12 days
  Firmness after one bite will be rated on a 100-mm VAS scale ranging from 'not at all' to 'extremely' with anchors at the beginning and end of the line
Thickness | Two periods of 12 days
  Thickness after one bite will be rated on a 100-mm VAS scale ranging from 'not at all' to 'extremely' with anchors at the beginning and end of the line
Chewiness | Two periods of 12 days
  Chewiness after one bite will be rated on a 100-mm VAS scale ranging from 'not at all' to 'extremely' with anchors at the beginning and end of the line
Dryness | Two periods of 12 days
  Dryness after one bite will be rated on a 100-mm VAS scale ranging from 'not at all' to 'extremely' with anchors at the beginning and end of the line
Cohesiveness | Two periods of 12 days
  Cohesiveness after one bite will be rated on a 100-mm VAS scale ranging from 'not at all' to 'extremely' with anchors at the beginning and end of the line
Elasticity | Two periods of 12 days
  Elasticity after one bite will be rated on a 100-mm VAS scale ranging from 'not at all' to 'extremely' with anchors at the beginning and end of the line
Springiness | Two periods of 12 days
  Springiness after one bite will be rated on a 100-mm VAS scale ranging from 'not at all' to 'extremely' with anchors at the beginning and end of the line
Stickiness | Two periods of 12 days
  Stickiness after one bite will be rated on a 100-mm VAS scale ranging from 'not at all' to 'extremely' with anchors at the beginning and end of the line
Familiarity | Two periods of 12 days
  Familiarity (after one bite and after the meal) will be rated on a 100-mm VAS scale ranging from 'not at all' to 'extremely' with anchors at the beginning and end of the line
Expected satiation | Two periods of 12 days
  Expected satiation (after one bite) will be rated on a 100-mm VAS scale ranging from 'not at all' to 'extremely' with anchors at the beginning and end of the line
Desire to eat the meal | Two periods of 12 days
  Desire to eat the meal (after one bite and after the meal) will be rated on a 100-mm VAS scale ranging from 'not at all' to 'extremely' with anchors at the beginning and end of the line
Reasons for eating cessation | Two periods of 12 days
  Reasons for eating cessation assessed with the Reasons Individuals Stop Eating Questionnaire (RISE-Q)
Eating rate (g/min) | Two periods of 12 days
  Eating rate (g/min) measured with video recording and automated video analysis
Number of chews (chews/gram and chewes/bite) | Two periods of 12 days
  Number of chews measured with video recording and automated video analysis
Number of bites | Two periods of 12 days
  Number of bites measured with video recording and automated video analysis
Bite size | Two periods of 12 days
  Bite size (gram/bite) measured with video recording and automated video analysis
Oral processing duration (minutes) | Two periods of 12 days
  Oral processing duration (minutes) measured with video recording and automated video analysis
Oro-sensory exposure time (s/g) | Two periods of 12 days
  Oro-sensory exposure time (s/g) measured with video recording and automated video analysis
Physical activity | Two periods of 12 days
  Energy expenditure will be measured using ActiGraph activity monitors
Energy expenditure | Two periods of 12 days
  Physical activity will be measured using ActiGraph activity monitors
Energy intake during wash-out period | Period of 16 days
  Energy (kcal) measured with a food dairy during the wash-out period
Macro-nutrient intake during wash-out period | Period of 16 days
  Macro-nutrient intake (g) measured with a food dairy during the wash-out period
Ultra-processed food intake during wash-out period | Period of 16 days
  UPF intake (%) measured with a food dairy during the wash-out period
Habitual energy intake | One hour
  Energy (kcal) measured with a food frequency questionnaire
Habitual macro-nutrient intake | One hour
  Macro-nutrient (g) measured with a food frequency questionnaire
Habitual ultra-processed food intake | One hour
  UPF intake (%) measured with a food frequency questionnaire
Habitual physical activity | Ten minutes
  Habitual physical activity (MET-min/week) measured using the short version of the International Physical Activity Questionnaire (IPAQ)
Habitual energy expenditure | Ten minutes
  Habitual energy expenditure (kcal/week) measured using the short version of the International Physical Activity Questionnaire (IPAQ)
Self-reported eating rate | One minute
  Self-reported eating rate measured using the question "How would you describe your eating rate compared with others?" which can be answered on a five-point Likert scale ('very slow', 'slow', 'average', 'fast' or 'very fast')
Restrained eating, emotional eating and external eating | Thirty minutes
  The level of restrained, emotional, and external eating assessed with the Dutch Eating Behaviour Questionnaire (DEBQ) consisting out of 33 questions.
Diet satisfaction | Ten minutes
  The Diet Satisfaction Questionnaire (DSat-28) consists out of five scales accessed by 28 statements about the characteristics of the lifestyle and attitudes of individuals that reflect satisfaction within the diets
Appetitive traits | Ten minutes
  The Adult Eating Behaviour Questionnaire (AEBQ) will be used to characterize the appetitive traits of the participants (Hunot et al., 2016). The questionnaire consists out of 35 statements which can be scored from "Strongly agree" (1) to 'Strongly disagree" (5). The statements are summarized into the scales 'Enjoyment of food', 'Emotional over-eating', 'emotional under-eating', 'Food fussiness', 'Food responsiveness', 'Hunger', 'Slowness in eating', and 'Satiety responsiveness'.

CONTACTS AND LOCATIONS:
Locations (1):
- Wageningen University, Human Nutrition Department, Wageningen, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: No